CLINICAL TRIAL: NCT04133428
Title: Prospective Observational Study of the Sacubitril-Valsartan Treatment Effectiveness.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: FIS-SAC-2018-01
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2019-10

CONDITIONS: Heart Failure
Keywords: Heart failure; Severe systolic disfunction; Sacubitril-Valsartan
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sacubitril-Valsartan cohort: Patients with severe systolic disfunction (left ventricle ejection fraction<40%) heart failure that remain functional class II, III or IV after at least 3 months of optimal treatment and after being evaluated by the cardiologist by doing an echocardiography, blood test and clinical evaluation, start Sacubitril-Valsartan treatment.
  Interventions: Drug: Sacubitril-Valsartan

INTERVENTIONS:
Drug: Sacubitril-Valsartan — Evaluation of the Sacubitril-Valsartan treatment effectiveness.
  As there are three possible doses, during the first 30 days of treatment 3 evaluations will be carried out (every 10 days) for dose titration based on safety and tolerability as well as a blood test the 30rd day of treatment.
  Afterwards the patient will be evaluated after 3 and 6 months of treatment with a blood test and in the final visit (6 months) an echocardiography will be carried out and the final clinical evaluation will be made.

SUMMARY:
The aim of this prospective study is to demonstrate if there is any difference in the treatment response to Sacubitril-Valsartan depending on the ventricular disfunction ethiology in patients with severe systolic disfunction heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old.
* Ejection fraction (EF) ≤ 40%.
* Treated with optimal medical treatment for at least 3 months and remained in functional class II, III or IV.
* Patients with ischemic or non ischemic etiology.

Exclusion Criteria:

* Patients with enolic etiology.
* Patients with any contraindication for taking Sacubitril-Valsartan.
* Patients with EF >40%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years old, diagnosed with heart failure and EF ≤ 40%, that after being treated with optimal medical treatment for at least 3 months, remain in functional class II, III or IV. Being this the actual indication for Sacubitril-Valsartan.
  100 consecutive patients will be included, 50 of whom with ischemic etiology of heart failure and 50 with non-ischemic, excluding patients with enolic etiology, any contraindication for the treatment intake and that have already been treated with Sacubitril-Valsartan.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-04-04 (Actual); Primary Completion 2021-04-04 (Estimated); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
Difference in the treatment response to Sacubitril-Valsartan depending on the ventricular dysfunction etiology. | Up to 6 months after the beginning of the Sacubitril-Valsartan treatment
  Verify if there is any difference in the response to the treatment with Sacubitril-Valsartan depending on the ventricular dysfunction etiology, ischemic or non-ischemic (idiopathic/familiar,toxic, volume overload,etc) excluding enolic, of patients with severe systolic heart failure.

SECONDARY OUTCOMES:
Determine the microRNA genetic profile in heart failure. | Up to 6 months after the beginning of the Sacubitril-Valsartan treatment
  Study of the microRNA genetic profile in heart failure as an indicator of the cardiac remodeling process and see its response and changes after undergoing Sacubitril-Valsartan treatment.

OTHER OUTCOMES:
Evaluate the connection between the biomarkers levels in heart failure and the cardiac remodeling parameters. | Up to 6 months after the beginning of the Sacubitril-Valsartan treatment
  Demonstrate if there´s a possible relation between the biomarkers levels in heart failure and an improvement in the cardiac remodeling.
Study the levels of auricular natriuretic peptide (ANP), auricular natriuretic peptide type B (BNP), urocortin and type I-C terminal pro-collagen. | Up to 6 months after the beginning of the Sacubitril-Valsartan treatment
  Study the levels of ANP, BNP and urocortin as cardioprotective molecules as well as type I-C terminal pro-collagen as measurement of peripheral blood fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Baron Esquivias, Principal Investigator — Hospital Universitario Virgen Macarena
Locations (1):
- Hospital Universitario Virgen Rocío, Seville, Spain